CLINICAL TRIAL: NCT04807374
Title: Use of a Hybrid Closed Loop Insulin Delivery System in a High Risk Type 1 Diabetes Population
Brief Title: Hybrid Closed Loop in High Risk Youth With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Tandem Diabetes Care, Inc. (Industry); DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Amanda Perkins, Adv Pract Nurse Practitioner, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013963
Record Dates: First submitted 2021-03-11; First posted 2021-03-19 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Type 1 Diabetes
Keywords: hybrid closed loop insulin delivery; healthcare disparities; diabetes technology
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: non-randomized interrupted time series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single arm- HCL Therapy (Experimental): Single arm study with all participants being treated with HCL for 6 months given the non-randomized interrupted time series study design.
  Interventions: Device: Control IQ

INTERVENTIONS:
Device: Control IQ — We aim to conduct a non-randomized prospective interrupted time series pilot study to investigate the effect of HCL insulin delivery on glycemic control in underserved adolescents with poorly controlled T1D.

SUMMARY:
The use of insulin pumps and continuous glucose monitors for Type 1 diabetes (T1D) has been shown to improve glycemic control while also decreasing the risk for acute and chronic complications. Unfortunately, there are vast disparities in access to this technology; non-Hispanic black youth with public healthcare insurance are the least likely to have access to these technologies. We propose to conduct a non-randomized interrupted time series study to assess the impact of hybrid closed loop (HCL) insulin delivery in underserved youths with poorly controlled T1D. Patients will complete standard diabetes education before beginning to use this technology and will be followed for 6-months after starting HCL to assess its impact on glycemic control and health-related quality of life.

DETAILED DESCRIPTION:
T1D is among the most common chronic childhood illness, affecting an estimated 1 in 400 American children.2 The care of children and adolescents with type 1 diabetes aims to optimize glycemic control to prevent acute and chronic complications of both hypoglycemia and hyperglycemia.

CGMs are minimally invasive devices that use a subcutaneous sensor to report and record changes in interstitial glucose values every 5 minutes to 15 minutes.6 This technology can alert patients to hypoglycemia and hyperglycemia and also allows them to make diabetes treatment decisions without the need for a confirmatory fingerstick blood glucose level. Improvements in the accuracy and usability of CGM, better insurance coverage, and greater acceptance by both clinicians and patients have led to dramatic increases in the use of this technology over the past decade.1,7-15 In 2011, just 6% of all patients in the United States Type 1 Diabetes Exchange (T1DX) registry were using CGM as compared to 27% in the period from 2016-2018.1 The use of CGM therapy has been associated with decreased hypoglycemia and severe hypoglycemia,16,17 improvements in A1c,1 reduced fear of hypoglycemia,18 and improved diabetes treatment satisfaction.19 Insulin pump therapy provides a continuous subcutaneous infusion of rapid acting insulin that allows for more physiologic insulin delivery as compared to multiple daily injection therapy. The use of insulin pump therapy in children with T1D has been associated with improved glycemic control, decreased rates of DKA, lower risk for microvascular complications, as well as psychosocial benefits.

Recently, input from CGM has been used to guide automated insulin delivery through insulin pumps in what is referred to as HCL insulin delivery. The Control IQ algorithm developed by Tandem Diabetes Care, Inc. uses a Dexcom G6 to adjust insulin delivery according to predicted glucose levels in 30 minutes to maximize TIR. Control IQ was FDA approved for patients with T1D ≥ 14 years of age in December 2019 and for patients ≥ 6 years of age in June 2020. A 6-month randomized controlled study of the Control IQ algorithm showed improvements in mean glucose, TIR, time in hypoglycemia, and time in hyperglycemia.25 Although Control IQ was shown to have positive impacts on glycemic control, its impact on those in poor glycemic control remains largely unknown. Prior studies included only a selected population: 86% of participants were white, 86% of participants had at least a bachelor's degree, 62% had an annual household income >$100,000, and the average A1c on enrollment was 7.4 ± 1.0%.

The increasing use of insulin pumps and continuous glucose monitors (CGM) among people with Type 1 diabetes (T1D) has been associated with worsening already existing healthcare disparities among people of different races, ethnicities, and socioeconomic statuses. Studies have shown that CGM use is more likely among participants with higher household incomes, greater levels of parental education, and those with private healthcare insurance.8 The disparities in access to these technologies persist even after controlling for these factors, which raises concern for clinician bias in prescribing these technologies despite evidence from an RCT that CGM use is equally beneficial for children of different racial and ethnic groups.26 There has been an ongoing push to better understand the various factors contributing to these disparities in access to diabetes technologies.27 Evidence that technology use varies according to geographic location speaks to the role of provider preference as well as patient socioeconomic status.28 The association between black race and higher rates of DKA and mortality in patients with T1D <25 years of age may impact provider insulin pump prescribing practices.29 While ongoing work is necessary to better understand factors impacting prescribing practices, the addition of data supporting the effectiveness of HCL therapy without higher rates of DKA in underserved patients can only help to strengthen this argument.

We aim to explore the effect of HCL insulin therapy with the Control IQ system on glycemic control as measured by time in range (TIR) in underserved youths ≥ 6 to < 21 years of age with poorly controlled T1D. For the purposes of this study, because of the lowest rates of diabetes technology use in this group, underserved patients will be defined as: non-Hispanic black with public healthcare insurance being managed with insulin regimens using either NPH or sliding scales. Poorly controlled T1D will be defined as: at least two A1c values ≥10% in the preceding year. We have specifically chosen these inclusion criteria for the purposes of this pilot study because we wish to show the effectiveness of using these technologies in patients who are the least likely to have access to diabetes technologies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients clinically diagnosed with T1D managed with insulin for at least 1 year
2. Black race
3. Public healthcare insurance
4. Male or female ages ≥ 6 and < 21 years
5. Not currently using insulin pump therapy
6. Poorly controlled T1D: one A1c value ≥ 10% in the preceding two years and a second A1c value ≥ 10% at enrollment
7. Investigators and primary clinical endocrine clinician have confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol
8. Living with one or more parent/legal guardian/ friend (for adults only) knowledgeable about emergency procedures for severe hypoglycemia and able to contact the participant in case of an emergency.
9. Total daily insulin dose of at least 10 units per day based on FDA approval for Control IQ
10. For females, not currently known to be pregnant If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of child-bearing potential at study entry and can be repeated as necessary in case of clinical concern. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
11. Not currently using and willingness not to start any non-insulin glucose-lowering agent during the course of the trial
12. Fluent in English as the Control IQ technology is currently available only in English
13. Willing to adhere to the study regimen

Exclusion Criteria:

1. Concurrent use of any non-insulin diabetes medications
2. More than 3 episodes of DKA in the year prior to enrollment
3. Major illnesses other than T1D
4. Significant cognitive limitations and major psychiatric disorders
5. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk
6. Participation in another pharmaceutical or device trial at the time of enrollment or during the study
7. Having immediate family members employed by Tandem Diabetes Care, Inc., TypeZero Technologies, LLC, Dexcom, Inc. or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Change in CGM Time in Range (TIR) | 6 months
  To explore the effect of HCL insulin therapy with the Control IQ system on glycemic control as measured by time in range (TIR) in underserved youth with poorly controlled T1D.

SECONDARY OUTCOMES:
Changes in mean CGM glucose | 6 months
Changes in glycemic management indicator (GMI) | 6 months
Changes in coefficient of variation of mean glucose | 6 months
Changes in CGM time in hypoglycemia (<70 mg/dL) | 6 months
Changes in CGM time in hyperglycemia (>180 mg/dL) | 6 months
Glycemic control as measured by hemoglobin A1c | 6 months
Incidence of diabetic ketoacidosis (DKA) | 6 months
Incidence of severe hypoglycemia | 6 months
Incidence of emergency department visits and hospital admissions | 6 months
Changes in youth perceptions of diabetes-specific quality of life | 6 months
  As measured by Type 1 Diabetes and Life (T1DAL)
Changes in youth perceptions of diabetes distress | 6 months
  As measured by Problem Areas in Diabetes (PAID)
Changes in youth perceptions of automated insulin delivery systems | 6 months
  As measured by INsulin Dosing Systems: Perceptions, Ideas, Reflections, and Expectations (INSPIRE)
Changes in youth perceptions diabetes self-management | 6 months
  As measured by Diabetes Management Questionnaire (DMQ)
Changes in youth attitudes about diabetes technologies | 6 months
  As measured by Diabetes Technology Attitudes Survey (DTAS)
Changes in parental perceptions of the youth's diabetes-specific quality of life | 6 months
  As measured by Type 1 Diabetes and Life (T1DAL) for Parents of People with Type 1 Diabetes
Changes in parental perceptions of the youth's diabetes distress | 6 months
  As measured by Parent Problem Areas in Diabetes (PAID)
Changes in parental perceptions of the youth's perceptions of automated insulin delivery systems | 6 months
  As measured by INsulin Dosing Systems: Perceptions, Ideas, Reflections, and Expectations (INSPIRE)
Changes in parental perceptions of the youth's diabetes management | 6 months
  As measured by Diabetes Management Questionnaire (DMQ) for parents
Changes in parental perceptions of the youth's attitudes about diabetes technologies | 6 months
  As measured by Parent Diabetes Technology Attitudes Survey (DTAS)
Semi-structured interviews with youth and parents exploring the overall experience and barriers to expanding access to hybrid closed loop technology | Post-Intervention at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Perkins, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marks BE, Grundman JB, Meighan S, Monaghan M, Streisand R, Perkins A. Hybrid Closed Loop Systems Improve Glycemic Control and Quality of Life in Historically Minoritized Youth with Diabetes. Diabetes Technol Ther. 2024 Mar;26(3):167-175. doi: 10.1089/dia.2023.0450. PMID 38444316